CLINICAL TRIAL: NCT02278783
Title: Phase 2 Trial of Regorafenib in Patients With Recurrent Ovarian, Primary Peritoneal and Fallopian Tube Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: University of Utah (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI77685
Record Dates: First submitted 2014-10-23; First posted 2014-10-30 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib Treatment arm, all patients (Experimental)
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — Patients will be treated with Regorafenib 160 mg (4 x 40 mg tablets) daily for 21 days of a 28 day cycle (three weeks on drug, one week off) until disease progression or adverse effects prohibit further treatment

SUMMARY:
This will be a non-blinded, single arm study to test the efficacy of Regorafenib in patients with recurrent ovarian, primary peritoneal, and fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

Age greater than or equal to 18 years. Life expectancy of at least 12 weeks (3 months). Diagnosis of recurrent epithelial ovarian, primary peritoneal or fallopian tube cancer. Histologic or cytologic confirmation of the original primary tumor is required.

Patients must have measurable disease defined as at least one lesion that can be accurately measured in at least one dimension with longest diameter (LD) greater than or equal to 10 mm using CT, MRI, or caliper measurements or greater than or equal to 20 mm with x-ray.

Patients must have at least one target lesion to be used to assess response on this protocol as defined by RECIST 1.1.

Prior therapy: Patients must have had at least one prior platinum-based chemotherapeutic regimen for management of primary disease containing Carboplatin, Cisplatin, or another organo-platinum compound. This initial treatment may have included intraperitoneal therapy, consolidation, non-cytotoxic agents (including anti-angiogenesis agents) or extended therapy (i.e. maintenance therapy) administered after surgical or non-surgical assessment.

Patients are allowed to have previously received, but are not required to receive, one or two additional cytotoxic regimens for management of recurrent disease.

Patients who have received only one prior cytotoxic regimen (platinum based regimen for management of primary disease), must have a platinum-free interval of at least 6 months.

Patients must not have received any non-cytotoxic therapy for management of recurrent or persistent disease, except hormonal based therapy is allowed. Patients are allowed to have previously received, but are not required to have received non-cytotoxic therapy as part of their primary treatment regimen.

ECOG score of 0-1. Adequate bone marrow, liver and renal function

Exclusion Criteria:

Patients who have progressed during initial platinum-based therapy in the upfront setting, who have persistent disease after this initial platinum-based therapy, or who have recurrence less than 6 months from adjuvant chemotherapy are excluded.

Major surgical procedure or significant traumatic injury within 28 days before start of study medication.

Patients who have received wide field radiotherapy less than or equal to 4 weeks or limited field radiation for palliation less than or equal to 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) greater than or equal to 5 effective half-lives prior to starting study drug or who have not recovered from side effects of such therapy.

Patients who have received chemotherapy or targeted anticancer therapy greater than or equal to 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C, and 1 week for hormone therapy) prior to starting study drug or who have not recovered from side effects of such therapy.

Active concurrent primary malignancy or prior malignancies occurring within 3 years (except cervical carcinoma in-situ, treated basal cell carcinoma, or superficial bladder tumor.

Use of any investigational drugs, biologics, or devices within 28 days prior to study enrollment.

Prior use of regorafenib. Strong inducers and inhibitors of CYP3A4 and therapeutic anticoagulation with Vitamin-K antagonists (e.g. warfarin) or with heparins and heparinoids Women who are pregnant or breastfeeding. Uncontrolled hypertension defined as systolic pressure greater than or equal to 140 mmHg or diastolic pressure greater than or equal to 90 mmHg despite optimal medical management.

Human immunodeficiency virus (HIV) positive diagnosis with a CD4 count of <100 mm3 or detectable viral load within the past 3 months, and is receiving combination anti-retroviral therapy.

Active or clinically significant cardiac disease Evidence or history of bleeding diathesis or coagulopathy Any hemorrhage or bleeding event ≥ NCI CTCAE v4.0 Grade 3 within 4 weeks prior to start of study medication.

Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment.

Patients with pheochromocytoma Symptomatic metastatic brain or meningeal tumors. Ongoing infection Presence of a non-healing wound, non-healing ulcer, or bone fracture Patient's with a history of kidney disease or persistent proteinuria must have less than Grade 3 proteinuria per NCI CTCAE v4.0 at screening.

Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.

Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 71 [71 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival (PFS)
Description: To evaluate the anti-tumor activity of Regorafenib as measured by progression free survival at 6 months in patients with recurrent gynecological cancers
Time Frame: Patients will be checked for PFS after 6 months on treatment
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1
participants | 1

2. Primary Outcome: Incidence of Adverse Events (Grade 2 or Higher), Assessed According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Description: To determine the nature and degree of toxicity of Regorafenib in this cohort of patients. Toxicity will be summarized by attribution: regorafenib-related adverse events grade 2 or higher will be reported.
Time Frame: Patients will remain on treatment for approximately 4-6 months on average.
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 1
participants | 1

3. Secondary Outcome: Estimate Progression Free Survival
Description: To estimate progression free survival for patients treated with this regimen
Time Frame: At 6 months patients will be checked for PFS, and compared to the expected probability of the patient being alive and progression-free for at least 6 months
Population: Study was terminated early, no analysis performed.
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Frequency of Clinical Benefit (Stable Disease, Partial and Complete Response)
Description: To determine the frequency of clinical benefit (stable disease, partial, and complete response) according to RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 criteria
Time Frame: Scans will be done every 2 cycles (every 2 months) for disease assessment. Patients on average will be on treatment for 4-6 months
Population: Study was terminated early, no analysis performed.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=1)
anemia (Blood and lymphatic system disorders) | 1
tachycardia (Cardiac disorders) | 1
oral mucositis (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
chills (General disorders) | 1
platelet count decrease (Investigations) | 1
creatinine increased (Investigations) | 1
AST increased (Investigations) | 1
weight loss (Investigations) | 1
hyponatremia (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
headache (Nervous system disorders) | 1
dizziness (Nervous system disorders) | 1
hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
palmar-plantar eythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
macular rash (Skin and subcutaneous tissue disorders) | 1
hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No